CLINICAL TRIAL: NCT05970237
Title: A Multicenter, Prospective, Non-interventional, Observational Study to Evaluate the Efficacy and Safety of Dapagliflozin in Patient With Type 2 Diabetes Mellitus and Hypertension
Brief Title: A Study to Evaluate the Efficacy and Safety of Dapagliflozin in Patient With Type 2 Diabetes Mellitus and Hypertension
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-DGF-OS-401
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of dapagliflozin in patient with type 2 diabetes mellitus and hypertension

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with type 2 diabetes mellitus accompanied by hypertension who are scheduled to be administrated Trudapa Tab. or Trudapa M SR Tab.
* Those who voluntarily signed a written personal information agreement to participate in this clinical study.
* Those able to understand this study, be cooperative in the execution of the study, and participate in the study until its completion.

Exclusion Criteria:

* Patients with secondary hypertension: Secondary hypertension is not limited to the following diseases; (e.g., coarctation of the aorta, hyperaldosteronism, renal artery stenosis, pheochromocytoma, Cushing's syndrome and polycystic kidney disease, etc.)
* Those who have a history of taking dapagliflozin within 4 weeks of baseline (Visit 1)
* Those who are expected to need insulin prescription during the study period
* Pregnant women, breast-feeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus accompanied by hypertension who are scheduled to be administrated Trudapa Tab. or Trudapa M SR Tab.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-10-21 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Target blood pressure control rate | 12weeks after administration
Target blood glucose achievement rate | 12weeks after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, Namdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No